CLINICAL TRIAL: NCT01626339
Title: Effect of Intravitreal Anti-Vascular Endothelial Growth Factors on Retinal Vessels Diameter
Brief Title: Effect of Intravitreal Anti-VEGF on Retinal Vessels Diameter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Other Study IDs: PPUM/MDU/300/04/03
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Age Related Macular Degeneration
Keywords: Anti vascular endothelial growth factor; retinal vessels
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Intravitreal Ranibizumab
  Other Names: Lucentis
Drug: Intravitreal bevacizumab
  Other Names: Avastin

SUMMARY:
Patients who will be scheduled for intravitreal injection of Ranibizumab or Bevacizumab will be recruited in this prospective self-controlled trial. Fundus photography will carried out at baseline immediately before injection and at 3, 7 days and 30 days after the first injection. Using image analysis software, measurements summarized as the central retinal artery equivalent (CRAE) and central retinal vein equivalent (CRVE).

Null Hypothesis: There is no significant difference between arteriolar/venular diameter before and after injection of intravitreal ranibizumab/bevacizumab in the treated and untreated eye

ELIGIBILITY:
Inclusion Criteria:

• Patients who wish and need bevacizumab or ranibizumab treatment for underlying disease

Exclusion Criteria:

* History of previous systemic or ocular Anti-VEGF therapy
* History of previous intravitreal injection with any drug
* Intraocular pressure ≥ 22
* Glaucoma
* History or presence of thromboembolic events
* Un-controlled blood pressure
* Blood donation during the previous 3 weeks
* Relevant media opacity of the lens

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Malaya Medical Center, Kuala Lumpur, Kuala Lumpur, Malaysia